CLINICAL TRIAL: NCT06944067
Title: Observational Study to Determine Red Blood Cell Alloimmunization Risk Etiology in Patients With Sickle Cell Disease
Brief Title: Study to Understand the Genetic Risk of Developing an Immune Response After Blood Transfusions Among Individuals With Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002264; 002264-HG
Record Dates: First submitted 2025-04-24; First posted 2025-04-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Transfusion; Alloimmunization
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alloimmune non-responders: Individuals with sickle cell disease who have received blood transfusions but never had an alloimmune response to transfusion.
- Alloimmune responders: Individuals with sickle cell disease who have a history of an alloimmune response when receiving blood transfusions.

SUMMARY:
The purpose of this research study is to look at genes and determine how they interact with each other to find changes that could explain why some people's immune systems may respond to blood transfusions. This response is called an alloimmune response. We strongly believe that when someone has an alloimmune response, it is caused by changes in their genes. We plan to compare changes in the genes of individuals that develop red blood cell alloimmunization after blood transfusions with those that do not develop alloimmunization. This may help us to create more targeted therapeutic interventions, which may improve the health of alloimmune responders.

DETAILED DESCRIPTION:
Study Description:

This study seeks to fine-map risk variants associated with increased susceptibility to developing red blood cell alloantibodies in patients with sickle cell disease (SCD), with the goal of characterizing the molecular basis of the alloimmunization response. This will allow for improved clinical management for individuals susceptible to alloimmunization responses.

Objectives:

Primary Objective:

Elucidate the role of previously identified risk loci in the development of alloantibodies among individuals with SCD.

Secondary Objective:

Validate and characterize additional, novel alloimmunization-related candidate loci.

Endpoints:

Primary Endpoint:

Completion of analysis of previously identified risk loci to determine the relationship between genome structure and expression.

Secondary Endpoint:

No additional candidate loci from concurrent discovery studies to evaluate.

ELIGIBILITY:
* INCLUSION CRITERIA

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Individual (> 2 years of age) with confirmed SCD diagnosis who meets at least one of the following conditions:

1. History of greater than ten administered transfusions or 20 transfusion units (where known)
2. History of one or more antibody screens
3. Known candidate variant genotype

EXCLUSION CRITERIA

An individual who meets any the following criteria will be excluded from participation in this study:

1. Impaired decision-making capability, with or without a legally authorized representative
2. History of transplant (e.g., organ, bone marrow, stem cell)
3. Taking immunosuppressive medications at time of enrollment
4. Confirmed pregnancy

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with sickle cell disease who may or may not have had a history of alloimmune response to blood transfusions. The study population will include children ages 2-17 years old and adults. The study population will not include pregnant women, people taking immunosuppressive medications, or people with a history of transplant (e.g., bone marrow or stem cell transplant).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2030-04-10 (Estimated); Study Completion 2030-04-10 (Estimated)

PRIMARY OUTCOMES:
Completion of analysis of previously identified risk loci to determine the relationship between genome structure and expression. | 5 years
  Analyze samples from study participants to determine whether they have the loci we previously identified.

SECONDARY OUTCOMES:
No additional candidate loci from concurrent discovery studies to evaluate. | 5 years
  When we can no longer identify new potentially causal loci, the study endpoint will be achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Hanchard, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002264-HG.html